CLINICAL TRIAL: NCT01124253
Title: Phase III Study of Adjuvant Vinorelbine Plus Cisplatin (NP) Versus NP Plus Endostar in Patients With Completely Resected Stage IB-IIIA Non-small Cell Lung Cancer
Brief Title: Adjuvant Vinorelbine Plus Cisplatin(NP) Versus NP Plus Endostar in Patients With Completely Resected Stage IB-IIIA Non-small Cell Lung Cancer(NSCLC)
Acronym: Dengshan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Municipal Science and Technology Commission (Other Government); Shanghai Chest Hospital (Other); Simcere Pharmaceutical Co., Ltd (Other)
Responsible Party: Meilin liao, shanghai chest hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: endo001
Record Dates: First submitted 2010-05-06; First posted 2010-05-17 (Estimated); Last update posted 2010-05-17 (Estimated); Status verified 2009-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: adjuvant therapy; non-small cell lung cancer; vinorelbine; cisplatin; recombinant human endostatin; endostar
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Endostatins; endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NP plus recombinant human endostatin (Experimental)
  Interventions: Drug: recombinant human endostatin
- vinorelbine plus cisplatin (No Intervention)
  Interventions: Drug: recombinant human endostatin

INTERVENTIONS:
Drug: recombinant human endostatin — recombinant human endostatin 15mg per ampul for injection 7.5mg/m2 IV (in the vein) on 1st to 14th days of a 21- day cycle, totally 4 cycles are needed
  Other Names: endostar

SUMMARY:
This study was designed to determine whether adjuvant vinorelbine plus cisplatin and endostar prolongs overall survival compare to vinorelbine plus cisplatin alone among patients with completely resected IB-IIIA non-small-cell lung cancer.

DETAILED DESCRIPTION:
It is an open labelled, randomized, mono-center phase III clinical trail.A total of 250 patients with resected stage IB to stage IIIA non-small cell lung cancer will either the group of vinorelbine plus cisplatin plus endostar or the group of vinorelbine plus cisplatin randomly. The primary end point was overall survival; principal secondary end points were recurrence-free survival and the toxicity and safety of the regimens.The major inclusive criteria are pathological confirmed non-small cell lung cancer after complete resection and can tolerate chemotherapy safely.The tissue and blood samples will be banked for further investigation. All of the enrolled patients will be followed up until death or over 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer, the pathology type includes squamous cell carcinoma, adenocarcinoma, large-cell carcinoma, and any mixed type of the 3 types mentioned above.
* Stage IB-IIIA non-small cell lung cancer, tumor was completely resected (The type of surgery including lobectomy, left side pneumonectomy,bi-lobectomy).
* The time from surgery to first dose of adjuvant chemotherapy are mandatory between 4-8 weeks.
* No evidence of tumor relapse prior to adjuvant therapy.
* Age 18-70, Eastern Cooperative Oncology Group(ECOG) performance status 0-1.
* Normal hematologic function.Renal function , hepatic and cardiac function will be within the acceptable ranges as following:serum bilirubin, aspartate aminotransferase(AST)and alamine aminotransferase(ALT)levels below 1.5 times of normal value.
* No history of chemotherapy or radiotherapy;
* The patient should have well compliance for chemotherapy and follow up
* Informed consent should be obtained before treatment.

Exclusion Criteria:

* The histological or cytological documents do not match the inclusion criteria.
* Right side pneumonectomy or any kind of incompletely resected surgery.
* The recruitment time are beyond 8 weeks from surgery.
* Any concurrent acute or chronic systemic diseases or psychiatric diseases, which might both increase the risks of the research itself or the medical therapy and influence the research results analysis. The researchers can make a judge for the following conditions to tell whether they are fit for this research:Uncontrolled high blood pressure, unstable angina , myocardial infarction , uncontrolled arrhythmia,or congestive heart failure with clinical symptoms within 12 weeks before randomization.Evidence of anemia from electrocardiographic manifestation or heart valve disease with confirmed clinical diagnosis.Clinically significant active infection state due to bacteria, virus and fungi invasion. Patients with grade II arrhythmia, grade II myocardial anemia, grade II abnormal cardiac troponin T, grade II high blood pressure or left ventricle ejection fraction (LVEF) less than 50 percent according to CTC 3.0 are not permitted to enrol the study.
* women with pregnant or lactation.
* Before enter the group,the patients had other malignant tumors except for non-melanoma skin cancer, carcinoma in situ and cured early-stage prostate cancer.
* With allergic constitution or possible allergic reflection to any known research drugs.
* Poor compliance.
* Not proper for the research according to the researchers' judgment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2007-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
overall survival(OS) | five years

SECONDARY OUTCOMES:
disease-free survival(DFS) | five years
the toxicity and safety | two years

CONTACTS AND LOCATIONS:
Overall Officials: Liao Meilin, M.D., Study Chair — Shanghai Chest Hospital; Lu sun, M.D., Study Director — Shanghai Chest Hospital
Locations (1):
- The Lung Cancer Center of shanghai chest Hospital, Shanghai, China

REFERENCES:
- [Derived] Zhou Z, Chen ZW, Yang XH, Shen L, Ai XH, Lu S, Luo QQ. Establishment of a biomarker model for predicting bone metastasis in resected stage III non-small cell lung cancer. J Exp Clin Cancer Res. 2012 Apr 26;31(1):34. doi: 10.1186/1756-9966-31-34. PMID 22537906